CLINICAL TRIAL: NCT07232836
Title: The Role of Cytokines and Neuroplasticity Modulators in the Development of Spinal Canal Stenosis and the Identification of Biomarkers for the Biochemical Evaluation of Treatment in Patients Undergoing Endoscopic Spinal Canal Decompression
Brief Title: Cytokines, Neuroplasticity Modulators, and Biomarkers in Spinal Canal Stenosis and Endoscopic Decompression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Collaborators: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Marzena Ratajczak, Principal Investigator, Poznan University of Physical Education
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PoznanUPhyEd no. 5
Record Dates: First submitted 2025-09-25; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Spinal Stenosis; Ligamentum Flavum Hypertrophy
Keywords: adipokines; biomarkers; endoscopic spinal canal decompression; inflammation; epidural adipose tissue
MeSH Terms: conditions — Spinal Stenosis; Inflammation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spinal Stenosis (Experimental)
  Interventions: Procedure: Endoscopic Spinal Canal Decompression
- No Spinal Stenosis (No Intervention): Tissues collected during surgery from people without spinal stenosis.
- No intervention (No Intervention)

INTERVENTIONS:
Procedure: Endoscopic Spinal Canal Decompression — Patients from the study group will undergo endoscopic decompression of the spinal canal, which involves the removal of tissues (bone, ligament, joint) causing compression of the neural structures of the spine and the possible removal of an abnormally displaced fragment of the intervertebral disc.
  Arms: Spinal Stenosis

SUMMARY:
Research Rationale and Study Design Lumbar spinal stenosis (LSS) is a common degenerative musculoskeletal disorder characterized by narrowing of the spinal canal, often leading to pain and disability. One of the primary contributors to this condition is hypertrophy (thickening) of the ligamentum flavum (LF), along with facet joint degeneration, intervertebral disc herniation, and ligament ossification. However, the pathophysiological mechanisms behind these changes remain incompletely understood.

Histological changes in hypertrophied LF include fibrocartilaginous metaplasia, type II collagen proliferation, ossification, calcium crystal deposition, and degeneration of elastic and collagen fibers. Both mechanical stress and inflammatory processes, particularly macrophage infiltration, are considered key contributors to degeneration, especially in the aging population. Yet, inflammation linked to systemic metabolic disorders-such as obesity and sarcopenia-may also significantly influence the degeneration of spinal structures.

Metabolic Inflammation and the Role of Adipokines Recent research has highlighted the role of adipokines in the pathogenesis of degenerative spinal and joint diseases. Disrupted lipid metabolism and chronic low-grade inflammation contribute to tissue remodeling, extracellular matrix (ECM) degradation, and ectopic fat deposition in spinal structures.

Epidural fat, normally present in the spinal canal, can become inflamed and secrete pro-inflammatory cytokines, potentially affecting adjacent tissues such as muscles and ligaments. Conditions like spinal epidural lipomatosis, which is associated with obesity, exemplify this pathological mechanism.

While adipokines like leptin and visfatin have been previously associated with LF ossification and degeneration, the presence and role of others-such as adipsin, vaspin, resistin, lipocalin-2, progranulin, chemerin, omentin-1, and GDF-15-have not yet been studied in LF or epidural fat. Given their known effects on inflammation and ECM remodeling, these molecules are strong candidates for involvement in spinal canal narrowing.

Research Hypotheses and Objectives

This study hypothesizes that adipose tissue-derived cytokines, particularly from epidural fat, contribute to LF degeneration and LSS through inflammatory and metabolic signaling. The main research objectives are to:

1. Identify differences in biomarker concentrations in LF, paraspinal muscle, and epidural fat from patients with and without LSS.
2. Determine correlations between tissue and blood biomarker levels and clinical parameters such as pain, disability, and body mass.
3. Select potential biomarkers for monitoring surgical outcomes of spinal decompression.
4. Identify cytokines that modulate LF inflammation and metabolism.
5. Evaluate the direct effects of adipokines on LF cell behavior in vitro. Study Design and Methods

   Study population:

   • 100 patients undergoing lumbar spine surgery at the Orthopaedic-Rehabilitation Clinical Hospital in Poznań:

   o 50 with LSS (ages 40-90)
   * 50 with disc herniation only (ages 18-40; control group)

   Tissue collection (intraoperative):

   • Ligamentum flavum

   • Paraspinal muscles

   • Epidural adipose tissue

   Blood samples:

   • Collected from all participants:

   o Within 48 hours before surgery

   o Two months post-surgery

   Clinical assessments:

   • Disability and pain scales
   * Preoperative MRI scans

   Laboratory analysis:

   • Molecular testing:
   * mRNA expression of selected cytokines and adipokines using PCR
   * Protein levels determined via ELISA in both serum and tissue homogenates • Cell culture studies:
   * One-third of collected tissue is used to establish primary cell cultures from LF, paraspinal muscles, and epidural fat
   * Cells will be stimulated with conditioned media from epidural fat and with selected recombinant cytokines (e.g., vaspin, lipocalin-2, GDF-15)
   * Experiments will assess the gene and protein expression of key molecules involved in inflammation, ECM remodeling, bone metabolism, fibrosis, and matrix degradation.

   The goal is to clarify the local and systemic roles of adipokines and inflammation in the pathogenesis of LF hypertrophy and LSS. This knowledge may aid in identifying biomarkers for disease progression and therapeutic targets for non-surgical interventions in the future.

DETAILED DESCRIPTION:
Spinal stenosis is a common musculoskeletal disorder that causes pain or disability in patients. However, the pathogenesis of this disease is complex and has not yet been fully elucidated. Lumbar spinal canal stenosis results from degenerative changes in structures located behind the spinal cord, such as hypertrophy of the ligamentum flavum (LF), as well as ligament calcification, degeneration and hypertrophy of the facet joints and/or herniation of intervertebral discs located anterior to the spinal cord. The pathology of LF hypertrophy includes fibrocartilaginous changes associated with type II collagen proliferation, ossification, calcium crystal deposition, degeneration of collagen and elastic fibers, and chondroid metaplasia of ligament fibroblasts. Numerous scientific studies have attempted to explore the etiology of hypertrophy and ossification of spinal ligaments, considering systemic, local, genetic, and environmental factors. However, the mechanism of degeneration development is still not fully understood. Besides mechanical stress and increased collagen synthesis (fibrosis) in the ligament, which make age a major risk factor, the presence of inflammation and macrophage infiltration is considered a significant contributor to degeneration development.

Therefore, it is reasonable to assume that the presence of inflammation associated with other health conditions-especially chronic ones-may, to an unknown extent, influence the course of spinal structure degeneration. Currently, obesity and sarcopenia are drawing particular attention as disorders affecting all systems of the human body. Since their prevalence is increasing, a thorough understanding of their consequences on individual organs has significant social and practical importance for prevention and health protection.

An increasing number of reports indicate that disturbances in lipid metabolism and the secretion of pro-inflammatory adipokines and cytokines are deeply involved in regulating cellular phenotypes and fates, extracellular matrix metabolism, and inflammation in the pathophysiological processes of degenerative spinal and joint diseases. Metabolic disorders can affect bone metabolism and lead to ectopic ossification and fat deposition not only in spinal ligaments but also in other spinal structures. Also noteworthy is the influence of the adipokinome on the development of musculoskeletal degenerative disorders. Even anatomically present epidural fat in the spinal canal may become inflamed and spontaneously secrete inflammatory cytokines, potentially modifying the function of adjacent tissues, such as paraspinal muscles and ligaments. It is worth mentioning that spinal epidural lipomatosis, characterized by an excess of fat tissue in the epidural space leading to spinal canal stenosis, is strongly associated with obesity.

So far, it has been confirmed that adipokines and their receptors, although primarily located in white adipose tissue, are also present in joint cartilage and spinal bone marrow. Adipokines may promote ligamentum flavum degeneration by stimulating inflammatory responses and promoting pathological changes. Leptin has been shown to significantly correlate with the number of vertebrae affected by ligamentous ossification. Fan et al. discovered that leptin markedly upregulates alkaline phosphatase and osteocalcin mRNA expression in ligamentum flavum cells. High levels of visfatin have also been found in the ligamenta flava of patients with confirmed ossification. There is no available data on the presence and role of other adipose tissue-derived cytokines such as adipsin, vaspin, resistin, lipocalin-2, progranulin, chemerin, omentin-1, or growth differentiation factor-15 (GDF-15) in the ligamentum flavum. It is highly likely that these cytokines are also involved in the development of spinal canal stenosis, which constitutes our research hypothesis. The presence and levels of these cytokines in epidural fat tissue in patients with stenosis, compared to those without spinal canal narrowing, have not been studied to date. Since studies confirm that chronic systemic inflammation affects various tissues and local inflammation significantly affects neighboring structures, we hypothesize that ligaments, paraspinal muscles, intervertebral discs, etc., may be particularly vulnerable to cytokines secreted by epidural fat tissue. Previous in vitro studies confirmed that a local environment rich in cytokines such as IL-6, IL-1α, nitric oxide donor (SNAP), and prostaglandin E2 changes the gene expression of collagens I, V, XI, and osteocalcin in ligamentum flavum cells. However, the impact of the mentioned adipokines on the development of ligamentum flavum degeneration has not yet been determined.

The study will involve examining the concentrations of cytokines (especially adipokines) and neuroplasticity modulators and their mRNA expression in tissues routinely removed from patients with spinal stenosis and disc herniation during surgery, as well as collecting blood from patients twice, before the procedure and during a follow-up visit two months after the procedure.

Objectives

1. To identify differences in selected biomarker concentrations in samples of ligamentum flavum, paraspinal muscles, and epidural fat collected from the lumbar region of patients with stenosis compared to those without spinal canal degeneration.
2. To determine whether the expression of selected biomarkers in tissues correlates with their presence in the patients' blood and whether they relate to the degree of degeneration, disability, pain intensity, and body mass.
3. To select potential biomarkers for monitoring the effectiveness of spinal canal decompression surgery by comparing biomarker levels before surgery and two months into recovery.
4. To identify potential proteins that modulate metabolism and inflammation in the ligamentum flavum.
5. To evaluate the impact of selected cytokines and adipokinome of epidural fat tissue on metabolism and inflammation in ligamentum flavum cell cultures.

Study Population Description

The study will involve 100 patients from the Orthopaedic-Rehabilitation Clinical Hospital of the Poznań University of Medical Sciences, including both men and women:

* 50 patients with lumbar spinal canal stenosis, aged 40-90 years
* 50 patients with intervertebral disc herniation, aged 18-40 years, requiring surgical treatment Participants will undergo surgery provided they give informed consent to use their tissues in scientific research.
* The study group will undergo endoscopic spinal canal decompression, involving the removal of tissues (bone, ligament, joint) compressing neural structures, and possibly removing a displaced intervertebral disc fragment.
* The control group will undergo isolated intervertebral disc herniation surgery, involving the removal of the displaced disc fragment.

Methods Before surgery (within 48h) and two months post-op, 20 ml of venous blood will be drawn from each patient.

During surgery, the following samples will be collected:

* Paraspinal muscle tissue
* Ligamentum flavum
* Epidural fat tissue

The study will use the following methods/tools:

1. Standardized questionnaires for disability and pain intensity
2. MRI of the lumbar spine (routinely performed before surgery)
3. Molecular testing

   1. mRNA expression of cytokines (GDF-15, adipsin, vaspin, resistin, lipocalin-2, progranulin, chemerin, omentin-1) will be measured using PCR.
   2. Immunoassays using commercial ELISA kits will be performed on tissue homogenates and serum to determine proteins concentrations (GDF-15, adipsin, vaspin, resistin, lipocalin-2, progranulin, chemerin, omentin-1)
4. Cell culture and stimulation of cells with cytokines and medium obtained from adipose tissue One-third of the biological material will be allocated for cell culture studies. Samples of the ligamentum flavum, paraspinal muscles, and epidural adipose tissue will be collected directly after surgery and placed in sterile containers with appropriate transport media.

All samples will be immediately transported to the cell culture laboratory under sterile conditions, in the shortest possible time from collection. Upon arrival at the laboratory, they will undergo appropriate, pre-established cell isolation protocols, tailored to the characteristics of each tissue type.

After the exposure period, the expression of mRNA and protein levels of cytokines, fibrosis markers, bone markers, extracellular matrix proteins, matrix degradation enzymes will be measured in the conditioned medium collected from the cultures of myocytes and ligamentum flavum fibroblasts.

ELIGIBILITY:
Inclusion Criteria for the experimental group:

1. Spinal stenosis in the lumbar spine with a referral for surgical treatment using endoscopic spinal decompression.
2. Age: 40-90 years.
3. Current MRI results.
4. Consent to participate in the study.

Inclusion Criteria for the control no spinal stenosis group:

1. Intervertebral disc herniation in the lumbar spine with a referral for surgical treatment using endoscopic discectomy.
2. Age: 18-40 years.
3. Current MRI results.
4. Consent to participate in the study.

Exclusion Criteria:

History of:

* rheumatoid arthritis of the intervertebral joints,
* joint pain located elsewhere if it is more severe than the pain caused by stenosis,
* pathologies and/or medications that may disturb the balance between pro- and anti-inflammatory factors (e.g. inflammatory diseases, rheumatoid arthritis, ankylosing spondylitis, acute infection),
* uncontrolled diabetes, poorly controlled hypertension, clinically significant liver function impairment, acute coronary event, unstable angina pectoris, symptoms of heart failure, pacemaker implantation,
* neurological diseases within the last 6 months,
* previous spine surgery at the lumbar level,
* mechanical injuries to the spine after an accident,
* advanced osteoporosis,
* pregnancy, lactation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-17 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Adipokines concentration in the epidural adipose tissue, paraspinal muscles, ligamentum flavum and blood. | Day 0 and Month 2
Neuroplasticity modulators concentration in the epidural adipose tissue, paraspinal muscles, ligamentum flavum and blood. | Day 0 and Month 2

SECONDARY OUTCOMES:
Low back pain on visual analogue scale | Day 0 and Month 2
  A horizontal or vertical line, 10 cm in length (0 to 10 scale) "0" represents "no pain" (or no symptom), and ten represents the "worst imaginable pain" (or most severe symptom).
Oswestry Disability Index | Day 0 and Month 2
  A self-reported questionnaire assessing how back pain affects a patient's ability to manage everyday life. The maximum score is 50 points, the minimum is 0. Higher scores mean worse outcome (more severe disability).
Thickness of the ligamentum flavum | Before intervention
  MRI
Diameter of the spinal canal | Before intervention.
  MRI
Schizas Scale | Before intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marzena Ratajczak, PhD, Principal Investigator — Poznan University of Physical Education

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Data will be available once the investigation is completed.
Access Criteria: Anonymised patient data may be transferred to the database in justified cases and at the request of the person concerned.

REFERENCES:
- [Background] Tarabeih N, Shalata A, Trofimov S, Kalinkovich A, Livshits G. Growth and differentiation factor 15 is a biomarker for low back pain-associated disability. Cytokine. 2019 May;117:8-14. doi: 10.1016/j.cyto.2019.01.011. Epub 2019 Feb 15. PMID 30776685
- [Background] Fujita N, Hosogane N, Hikata T, Iwanami A, Watanabe K, Shiono Y, Okada E, Ishikawa M, Tsuji T, Shimoda M, Horiuchi K, Nakamura M, Matsumoto M, Ishii K. Potential Involvement of Obesity-Associated Chronic Inflammation in the Pathogenesis of Idiopathic Spinal Epidural Lipomatosis. Spine (Phila Pa 1976). 2016 Dec 1;41(23):E1402-E1407. doi: 10.1097/BRS.0000000000001646. PMID 27105459
- [Background] Xiang Q, Wu Z, Zhao Y, Tian S, Lin J, Wang L, Jiang S, Sun Z, Li W. Cellular and molecular mechanisms underlying obesity in degenerative spine and joint diseases. Bone Res. 2024 Dec 11;12(1):71. doi: 10.1038/s41413-024-00388-8. PMID 39658574
- [Background] Endo T, Koike Y, Hisada Y, Fujita R, Suzuki R, Tanaka M, Tsujimoto T, Shimamura Y, Hasegawa Y, Kanayama M, Yamada K, Iwata A, Sudo H, Ishii M, Iwasaki N, Takahata M. Aggravation of Ossified Ligamentum Flavum Lesion Is Associated With the Degree of Obesity. Global Spine J. 2023 Jun;13(5):1325-1331. doi: 10.1177/21925682211031514. Epub 2021 Oct 6. PMID 34615403
- [Background] Zhang H, Hong Z, Jiang Z, Hu W, Hu J, Zhu R. miR-29b-3p Affects the Hypertrophy of Ligamentum Flavum in Lumbar Spinal Stenosis and its Mechanism. Biochem Genet. 2025 Apr;63(2):1824-1838. doi: 10.1007/s10528-024-10811-8. Epub 2024 Apr 16. PMID 38625592
- [Background] Furusawa N, Baba H, Maezawa Y, Uchida K, Wada M, Imura S, Fukuda M. Calcium crystal deposition in the ligamentum flavum of the lumbar spine. Clin Exp Rheumatol. 1997 Nov-Dec;15(6):641-7. PMID 9444420
- [Background] Szpalski M, Gunzburg R. Lumbar spinal stenosis in the elderly: an overview. Eur Spine J. 2003 Oct;12 Suppl 2(Suppl 2):S170-5. doi: 10.1007/s00586-003-0612-1. Epub 2003 Sep 9. PMID 13680315
- [Background] Silwal P, Nguyen-Thai AM, Alexander PG, Sowa GA, Vo NV, Lee JY. Cellular and Molecular Mechanisms of Hypertrophy of Ligamentum Flavum. Biomolecules. 2024 Oct 10;14(10):1277. doi: 10.3390/biom14101277. PMID 39456209
- [Background] Carregaro RL, Tottoli CR, Rodrigues DDS, Bosmans JE, da Silva EN, van Tulder M. Low back pain should be considered a health and research priority in Brazil: Lost productivity and healthcare costs between 2012 to 2016. PLoS One. 2020 Apr 1;15(4):e0230902. doi: 10.1371/journal.pone.0230902. eCollection 2020. PMID 32236113